CLINICAL TRIAL: NCT06434909
Title: An Investigator Sponsored Study to Investigate the Safety and Efficacy of CYTALUX™ (PAFOLACIANINE) INJECTION for the Intraoperative Imaging of Prostate Cancer
Brief Title: CYTALUX™for the Intraoperative Imaging of Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: On Target Laboratories, LLC (Industry)
Responsible Party: Principal Investigator, Clinton Bahler, Principal investigator, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IUSCCC-0890
Record Dates: First submitted 2024-05-17; First posted 2024-05-30 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: fluorescent; image guided intervention; folate; prostate cancer; laparoscopic prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pafolacianine; Surgery, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pafolacianine injection and surgery (Experimental)
  Interventions: Drug: Cytalux™ (pafolacianine) for fluorescent imaging; Procedure: Image Guided Surgery

INTERVENTIONS:
Drug: Cytalux™ (pafolacianine) for fluorescent imaging — Cytalux™ (pafolacianine) injection: folate analog ligand conjugated with an indole cyanine green-like dye for real-time cancer margin status.
  This is used in conjunction with appropriate imaging system.
Procedure: Image Guided Surgery — prostatectomy using appropriate imaging system

SUMMARY:
This study is being done to compare how much using Cytalux™ (pafolacianine) with NIR (Near InfraRed) fluorescent imaging improves the detection of malignant (growing in an uncontrolled way) tissue in adult subjects undergoing prostatectomy and lymph node dissection for biopsy confirmed prostate cancer.

The U.S. Food and Drug Administration (FDA) has approved the targeted imaging agent pafolacianine (Cytalux) for use in ovarian cancer (2021) and lung cancer surgery (2022.)

DETAILED DESCRIPTION:
This is an open label trial in up to 15 subjects with biopsy confirmed prostate cancer (PCa) who have been scheduled to undergo a laparoscopic radical prostatectomy with or without robotic assistance, with pelvic lymph node dissection. This is a non-intervention trial to assess the accuracy of an imaging agent, folate targeted fluorescent dye (pafolacianine), during a standard of care radical prostatectomy.

Qualifying subjects will be Grade Group 3 to 5 (>/= cT3) with either suspected extraprostatic disease (EPD) (extracapsular extension (ECE) and/or seminal vesicle infiltration (SVI)), or suspected lymph node metastasis (clinical stage cN1, or by magnetic resonance imaging (mriN+), or by Prostate Specific Membrane Antigen positron emission tomography (PSMA PET+).

Whether using an anterior or a posterior approach, the tissues planned for removal will be visualized first under normal light, and their locations marked on a provided template. All additional suspicious tissue or nodes will be similarly marked, whether removed or not. Prior to removal, the field must be illuminated with Near Infrared light (NIR) and fluorescent tissues must be marked on the template. This may proceed in an iterative fashion, switching from first normal light to NIR as the surgical field expands.

NIR imaging must be conducted in the timeframe of one hour to twenty-four hours following IV infusion of pafolacianine. Lymphatics to be examined are, at a minimum, the external iliac, internal iliac and obturator fossa, and common iliac. Fluorescence positive nodules and nodes will be removed at the surgeon's discretion and sent as labeled (specimen number, tissue, location) specimens to pathology without designation of florescence. Ink dots should ideally be applied to the spot suspected of being cancerous.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form and HIPAA form
2. Male subjects 18 years of age and older
3. Known primary prostate cancer
4. Grade Group 3 to 5 (≥cT3) with either:

   1. suspected extraprostatic disease (EPD) (extracapsular extension (ECE) and/or seminal vesicle infiltration (SVI)), or 3 or more biopsy cores of grade group 3-5;
   2. suspected lymph node metastasis (clinical stage cN1, or by magnetic resonance imaging (mriN+), or by Prostate Specific Membrane Antigen positron emission tomography (PSMA PET+));
   3. or both.
5. Planned to undergo a standard of care laparoscopic prostatectomy with or without robotic assistance, and lymph node dissection
6. Ability to understand the requirements of the study and agree to abide by the study restrictions and to return for the required assessments
7. Agree to stop folate or folic acid supplements at least 48 hours prior to injection of study agent

Exclusion Criteria:

1. The surgeon plans to perform an extraperitoneal approach
2. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the subject
3. History of anaphylactic reactions to products containing indocyanine green
4. History of allergy to any of the components of PAFOLACIANINE

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Detection of residual cancer | Day of surgery (visit 2)
  The proportion of subjects who have a Clinically Significant Event (CSE). A CSE is a composite endpoint defined as at least one of the following outcomes:
  1. One or more resected "NIR only" positive lymph nodes that contain metastatic disease as confirmed by pathology.
  2. Histologically confirmed cancer in resected "NIR only" residual non-nodal soft tissue following prostatectomy.

SECONDARY OUTCOMES:
Treatment change | Day of surgery (visit 2)
  To evaluate the proportion of subjects whose surgical procedure changed in scope from the planned surgery based on the use of PAFOLACIANINE with NIR imaging.
Differences in sensitivity and specificity of lesions | Day of surgery (visit 2)
  T evaluate proportion of lesions that are either: fluorescence positive, and prostate cancer positive; fluorescence positive but cancer negative; fluorescence negative but cancer positive; or, fluorescence negative and cancer negative.

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Bahler, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Health Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No